CLINICAL TRIAL: NCT02902887
Title: A Clinical Trial of Observation Versus Controlled Intermittent Alternate Occlusion (CIAO) Therapy for Intermittent Exotropia
Brief Title: Monitored Controlled Intermittent Alternate Occlusion (CIAO) Therapy for Intermittent Exotropia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Salus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HJW1601
Record Dates: First submitted 2016-05-08; First posted 2016-09-16 (Estimated); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Intermittent Exotropia
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Monitored CIAO therapy (Experimental): Participants wear 3-hour CIAO therapy
  Interventions: Device: Controlled Intermittent Alternate Occlusion (CIAO ) glasses
- Observation (No Intervention): No intervention, just observation

INTERVENTIONS:
Device: Controlled Intermittent Alternate Occlusion (CIAO ) glasses — Monitored CIAO therapy glasses
  Arms: Monitored CIAO therapy

SUMMARY:
This study presents an opportunity to understand a novel, previously unreported controlled intermittent alternate occlusion (CIAO) therapy glasses, which may improve the control of Intermittent exotropia (IXT).

ELIGIBILITY:
Inclusion Criteria:

The following criteria must be met for the patient to be enrolled in the study:

1. Age 3 to 11 years old
2. Intermittent exotropia (manifest deviation) meeting all of the following criteria:

   * Intermittent exotropia at distance OR constant exotropia at distance and either intermittent exotropia or exophoria at near
   * Exodeviation at least 10PD at distance OR 15PD at near measured by prism and alternate cover test (PACT)
3. No previous surgical or non-surgical treatment for IXT (other than refractive correction)
4. Visual acuity in the worse eye 20/40 (0.3 logMAR) or better on ATS HOTV for ages 3 - 5 and 20/25 (0.1 logMAR) or better on ATS HOTV for ages 6 - 11
5. No hyperopia greater than +3.50 D spherical equivalent in either eye
6. No myopia greater than -6.00 D spherical equivalent in either eye
7. Patients must be wearing refractive correction (spectacles or contact lenses) for at least one week if refractive error (based on cycloplegic refraction performed within 6 months) meets any of the following:

   * Myopia > -0.50 D spherical equivalent in either eye
   * Anisometropia > 1.00 D spherical equivalent
   * Astigmatism in either eye > 2.00 D if ≤ 5 years old and > 1.50 D if > 5 years old

   Refractive correction for patients meeting the above refractive error criteria must meet the following guidelines:
   * Anisometropia spherical equivalent must be within 0.25D of the full anisometropic difference correction
   * Astigmatism cylinder must be within 0.25D of full correction and axis must be within 5 degrees of full correction.
   * For hyperopia, the spherical component can be reduced at investigator discretion provided the reduction is symmetrical. Prescribing any refractive correction to yield lenses that are more myopic than -0.50 D spherical equivalent (SE) is considered deliberate overminus and is not allowed at enrollment. However, prescribing no correction or prescribing less than the full cycloplegic hyperopic correction (i.e., prescribing reduced plus) is not considered the same as overminusing for this protocol and is allowed because most patients without IXT but with hyperopic SE refractions in this range would not typically be prescribed a refractive correction.
   * For myopia, the intent is to fully correct, but the spherical component can be undercorrected by investigator discretion provided the reduction is symmetrical and results in no more than -0.50 D SE residual (i.e., uncorrected) myopia. Prescribing a correction that yields more than 0.50 D more minus SE than the cycloplegic refraction SE is considered deliberate overminus and is not allowed at enrollment.

   Note that the refractive correction guidelines and the requirement to wear refractive correction for at least one week apply not only to patients who require refractive correction under the above criteria but also to any other patient who is wearing refractive correction.
8. No atropine use within the last week
9. Gestational age > 34 weeks and birth weight > 1500 grams
10. Patient and/or parent is willing to accept randomization to either observation or CIAO therapy.
11. Parent has a phone (or access to phone) and is willing to be contacted

Exclusion Criteria:

1. Only phoria at both distance and near
2. Prior non-surgical treatment for IXT other than refractive correction (e.g., vergence therapy, occlusion, vision therapy/orthoptics, or deliberate over-minus with spectacles more than 0.50D)
3. Previous amblyopia treatment other than refractive correction within 1 year
4. Vision therapy/orthoptics for any reason within the last year
5. Interocular visual acuity difference more than 0.2 logMAR (2 lines on ATS HOTV for patients 3 to < 7 years old or 10 letters on E-ETDRS for patients ≥ 7 years old)
6. Investigator planning to initiate amblyopia treatment

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Control of the exodeviation assessment (scaled 1-5) | 3-month
  Intermittent Exotropia Control Scale (1-5) 5 = Constant exotropia 4 = Exotropia > 50% of the 30-second period before dissociation 3 = Exotropia < 50% of the 30-second period before dissociation 2 = No exotropia unless dissociated, recovers in > 5 seconds
  1 = No exotropia unless dissociated, recovers in 1-5 seconds 0 = No exotropia unless dissociated, recovers in < 1 second (phoria)

CONTACTS AND LOCATIONS:
Locations (1):
- Salus University, Elkins Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No